CLINICAL TRIAL: NCT02136654
Title: Novel Model for South Asian Treatment in Diabetes (NaMaSTe-Diabetes) Trial in Primary Care
Acronym: Namaste
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of British Columbia (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Khan, Professor, University of British Columbia
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Health Services Research
Other Study IDs: H14-00693
Record Dates: First submitted 2014-04-29; First posted 2014-05-13 (Estimated); Last update posted 2020-11-27 (Actual); Status verified 2020-11

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: diabetes; ethnicity; South Asian; diabetes management
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Culturally tailored diabetes program (Experimental): Culturally tailored diabetes program
  * culturally tailored diabetes education
  * lifestyle counselling
  * medication adherence counseling
  * peer supporter
  * communication training
  * family member involvement
  Interventions: Behavioral: Culturally tailored diabetes program
- Usual Care (No Intervention): Usual Care includes continuing to visit primary care physician for ongoing diabetes management Printed diabetes education materials.

INTERVENTIONS:
Behavioral: Culturally tailored diabetes program — Includes family member and peer support Includes communication training
  Arms: Culturally tailored diabetes program

SUMMARY:
South Asians (SA) living in Canada and globally have high rates of type 2 diabetes (diabetes). Despite the burden of diabetes in this population, diabetes management remains poor. SA patients are less likely to exercise, follow a healthy diet (4), participate in exercise programs (5), and are 24% less likely to achieve glucose, blood pressure and lipid targets for diabetes than the general population (6). 55-60% of SA patients were non-adherent to their diabetes life-saving medications, compared to 30-35% non-adherence in the general population (7). This large gap in diabetes care is not surprising given language and communication barriers between primary care providers and SA patients (8-10), lack of knowledge about diabetes (8-11), preference for alternative therapies (12-14) and fundamentally different cultural beliefs on diabetes and diabetes management (15-18). Although there is some preliminary evidence that culturally tailored, chronic disease models may improve outcomes (21-24), the current evidence base is insufficient to justify the system modifications required to provide culturally tailored care across primary care settings in Canada. We propose to conduct a randomized controlled trial to assess the impact of a novel culturally tailored lifestyle and medication adherence intervention in SA patients with poorly controlled diabetes. The study is called the Novel Model for South Asian diabetes Treatment (NaMaSTe-Diabetes) trial in primary care.

DETAILED DESCRIPTION:
South Asians living in Canada and globally have high rates of chronic diseases including hypertension, type 2 diabetes (diabetes) and cardiac disease (1-3). Diabetes is arguably one of the most pressing chronic diseases among South Asian (SA) populations as it occurs at 50% higher rates in SA patients than the general population, develops 5-10 years earlier, and is one of the principal causes of premature heart attack and death in this group (1). Despite the burden of diabetes in this population, diabetes management remains poor. Under the current health care system, SA patients are less likely to exercise, follow a healthy diet (4), participate in exercise programs (5), and are 24% less likely to achieve glucose, blood pressure and lipid targets for diabetes than the general population (6). 55-60% of SA patients were non-adherent to their diabetes life-saving medications, compared to 30-35% non-adherence in the general population (7). This large gap in diabetes care is not surprising given language and communication barriers between primary care providers and SA patients (8-10), lack of knowledge about diabetes (8-11), preference for alternative therapies (12-14) and fundamentally different cultural beliefs on diabetes and diabetes management (15-18). Although there is some preliminary evidence that culturally tailored, chronic disease models may improve outcomes (21-24), the current evidence base is insufficient to justify the system modifications required to provide culturally tailored care across primary care settings in Canada. We propose to conduct a randomized controlled trial to assess the impact of a novel culturally tailored lifestyle and medication adherence intervention in SA patients with poorly controlled diabetes. The study is called the Novel Model for South Asian diabetes Treatment (NaMaSTe-Diabetes) trial in primary care. The study aims to recruit 600 patients with type 2 diabetes and randomize them to either a culturally tailored lifestyle and medication adherence intervention (family based, culturally tailored diabetes self management education with ongoing peer support) versus usual care on glycemic control (change in A1C level) and change in blood pressure (systolic and diastolic blood pressure) from baseline to 6 months in SA patients with poorly controlled type 2 diabetes. The NaMaSTe trial is a multi-center individual randomized controlled trial of 600 SA patients with poorly controlled diabetes (A1C ≥7%) living in British Columbia, Canada.

ELIGIBILITY:
Inclusion Criteria:

* age >19 years of age
* type 2 diabetes mellitus requiring at least one medication (oral hypoglycemic agent and/or insulin) to control diabetes
* A1C ≥7% in past 1 year
* willingness/ability to attend the Diabetes education, dietician, and peer sessions and follow up assessments
* ability to provide informed consent
* self identify as South Asian (from India, Pakistan, Sri Lanka, or Bangladesh) regardless of generational status or timing of immigration with ability to speak in English or Punjabi.

Exclusion Criteria:

* life- limiting illness <12 months
* physical inability to exercise
* recurrent severe hypoglycemia or hypoglycaemic unawareness
* family member of, or living in same household as a participant
* pregnancy or gestational diabetes.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2015-07; Primary Completion 2021-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Change in A1C or blood pressure (systolic or diastolic blood pressure) | within 6 months from baseline; 0, 3, and 6 months

SECONDARY OUTCOMES:
change in fasting lipid profile | 6 months; 0 and 6 months
Change in weight or waist circumference | 6 months; 0, 3, and 6 months
change in health status | 6 months; 0, 3, and 6 months

OTHER OUTCOMES:
Procedure related outcomes | 6 months; 0, 3, and 6 months
  health behaviours, medication adherence, patient engagement/activation, diabetes management, diabetes distress, depression, social support, knowledge, motivation, self efficacy.

CONTACTS AND LOCATIONS:
Overall Officials: Nadia A Khan, MD MSc, Principal Investigator — University of British Columbia; Tricia Tang, PhD, Principal Investigator — University pf British Columbia
Locations (1):
- University of British Columbia, Vancouver, British Columbia, Canada